CLINICAL TRIAL: NCT07070960
Title: A Multicenter, Open-label, Single-arm Clinical Study of Anti-BCMA CAR-T Cell Therapy in Transplant-ineligible Patients With Newly Diagnosed Multiple Myeloma
Brief Title: A Study of Anti-BCMA CAR-T Therapy in Newly Diagnosed Myeloma Patients Who Are Transplant-ineligible
Acronym: CAR-T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, Chief Hematologist of The Affiliated Hospital of Xuzhou Medical University, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2025-KL280-01
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma; Newly Diagnosed
Keywords: Multiple Myeloma; transplant-ineligible; CAR-T
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T (Experimental): CAR-T alone
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — The T cells are genetically modified to express a chimeric antigen receptor targeting BCMA and are infused after induction therapy at a target dose of ≥2.0×10^6 cells/kg

SUMMARY:
This is a prospective study of anti-BCMA CAR-T in transplant-ineligible patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
After the diagnosis of multiple myeloma (MM), patients were stratified by frailty status. Frail patients received 4 cycles of VRd regimen (bortezomib, lenalidomide, and dexamethasone), while non-frail patients received 4 cycles of DVRd regimen (daratumumab, bortezomib, lenalidomide, and dexamethasone). Following induction therapy, peripheral blood lymphocytes were collected to manufacture anti-BCMA CAR-T cells. After lymphodepletion with the FC regimen (fludarabine and cyclophosphamide), patients received a single infusion of anti-BCMA CAR-T cells at a target dose of 2.0 × 10^6 CAR-positive cells per kilogram of body weight. Peripheral blood samples were collected at regular intervals to assess treatment efficacy, safety, and CAR-T cell expansion and persistence. Patients were closely monitored for 6 months post-infusion. Thereafter, disease assessments, physical examinations, and hematologic tests were conducted every 3 months for a total follow-up duration of 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years (inclusive);
2. Estimated life expectancy of more than 12 weeks;
3. Diagnosis of multiple myeloma confirmed by physical examination, pathological evaluation, laboratory tests, and imaging studies;
4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels less than 3 times the upper limit of normal (ULN);
5. Karnofsky Performance Status (KPS) score > 50%.
6. Ineligible for ASCT.

Exclusion Criteria:

1. Pregnant or lactating women, or women planning to become pregnant within the next six months;
2. Transduction efficiency of targeted lymphocytes <10%, or expansion fold <5× under CD3/CD28 co-stimulation, as determined by feasibility screening;
3. History of severe allergies or hypersensitivity, especially to interleukin-2 (IL-2);
4. Significant dysfunction of vital organs including the heart, lungs, or brain;
5. Any other condition that, in the investigator's judgment, makes the patient unsuitable for participation in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 36 months after CAR-T infusion
  Progression-Free Survival (PFS) is defined as the time from the date of CAR-T cell infusion to the date of disease progression or death from any cause, whichever occurs first. Disease progression will be determined based on the International Myeloma Working Group (IMWG) criteria. Patients who have not progressed or died will be censored at the date of last follow-up.
Overall Survival (OS) | Up to 36 months after CAR-T infusion
  Overall Survival (OS) is defined as the time from the date of CAR-T cell infusion to death from any cause. Patients who are alive at the time of analysis will be censored at their last known date of follow-up.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months after CAR-T infusion
  Objective Response Rate (ORR) is defined as the proportion of patients achieving a response of partial response (PR) or better, including PR, very good partial response (VGPR), complete response (CR), and stringent complete response (sCR), according to the International Myeloma Working Group (IMWG) criteria. The assessment will be based on laboratory parameters, imaging, and bone marrow evaluation, as applicable
MRD | Up to 36 months after CAR-T infusion
  The proportion and immunophenotype of plasma cells in bone marrow were analyzed using flow cytometry, with a sensitivity of 10^-5.
Adverse Events (AE) | Up to 36 months after CAR-T infusion
  Focus on adverse events related to ASCT and CAR-T, including CRS, ICANS, coagulation disorders, infections, and other complications。

CONTACTS AND LOCATIONS:
Overall Officials: Kailin Xu, Study Chair — The Affiliated Hospital oh Xuzhou Medical University

IPD SHARING:
Plan to Share IPD: No